CLINICAL TRIAL: NCT07297420
Title: Peri-Intubation Adverse Airway Events in Critically Ill Patients With Morbid and Super Obesity: A Retrospective Analysis
Brief Title: Peri-Intubation Adverse Airway Events in Critically Ill Patients With Morbid and Super Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: Zeliha Alicikus (Other Government)
Responsible Party: Sponsor-Investigator, Zeliha Alicikus, Head of Anesthesiology and Reanimation department,Assoc Prof, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: AYTEN-1
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Airway Complication of Anesthesia; Intubation; Difficult or Failed
MeSH Terms: conditions — Obesity | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Morbidly obese (BMI 40-49.9 kg/m²)
  Interventions: Procedure: endotracheal intubation
- Group 2: Super obese (BMI ≥50 kg/m²)
  Interventions: Procedure: endotracheal intubation

INTERVENTIONS:
Procedure: endotracheal intubation — adult trauma patients (≥18 years) admitted to the Surgical Intensive Care Unit

SUMMARY:
This study aims to compare the incidence and characteristics of peri-intubation adverse airway events in critically ill trauma patients with morbid obesity versus those with super obesity, and to determine whether increasing BMI independently predicts severe peri-intubation complications.

DETAILED DESCRIPTION:
Obesity represents a major global health challenge, with prevalence steadily rising worldwide. Beyond its well-characterized metabolic and cardiovascular consequences, obesity poses significant challenges for airway management, particularly among critically ill patients requiring urgent tracheal intubation. The degree of obesity is clinically relevant: morbid obesity (BMI ≥40 kg/m²) is associated with anatomical and physiological alterations that markedly increase the risk of difficult airway and peri-intubation complications compared with patients with BMI <40 kg/m².

From an anatomical perspective, morbidly obese patients often present with a short, thick neck, increased cervical adiposity, and limited atlanto-occipital extension, complicating optimal positioning and glottic visualization during laryngoscopy. Redundant upper airway soft tissue, macroglossia, and higher Mallampati classes further impede mask ventilation and reduce pharyngeal patency. Secondary analyses of the international INTUBE cohort demonstrated that obese critically ill patients had a significantly higher prevalence of difficult airway predictors such as short neck, reduced mouth opening, and high Mallampati scores, compared with non-obese patients (74.3% - 35.7%, p<0.001). Similarly, in a large retrospective bariatric cohort, severe obesity independently increased the odds of difficult intubation when Cormack-Lehane grade IV (OR 8.9) or Mallampati IV (OR 5.1) were present.

Physiological derangements further compound these challenges. Elevated intra-abdominal pressure and cephalad diaphragm displacement reduce functional residual capacity (FRC) and expiratory reserve volume, leaving critically limited oxygen reserves during apnea. Increased oxygen consumption and basal metabolic rate shorten the safe apneic window, resulting in rapid desaturation if intubation is prolonged or requires multiple attempts. The INTUBE study reported that severe peri-intubation hypoxemia (SpO₂ <80%) occurred more frequently in obese versus non-obese critically ill patients (12.1% - 8.6%, p=0.01), and first-pass intubation failure strongly correlated with this complication. Even in optimized elective settings such as bariatric surgery, BMI >60 kg/m² significantly increased the risk of difficult intubation, despite high first-pass success rates (95.4%) and low complication rates.

These findings highlight that morbid obesity imposes both anatomical and physiological barriers to safe intubation. Critically ill patients with morbid obesity are uniquely vulnerable, with increased risks of failed first-pass attempts, severe hypoxemia, and potentially life-threatening complications. However, prospective evidence directly comparing peri-intubation outcomes among critically ill patients with BMI 40-50 versus ≥50 kg/m² remains limited.

While morbid obesity is an established risk factor, there is a compelling physiological rationale to suspect heterogeneity of risk within this category. Super obesity (BMI ≥50 kg/m²) may represent a distinct phenotype with more pronounced anatomical and physiological derangements. In elective bariatric populations, BMI >50 kg/m² has been linked to difficult mask ventilation and intubation, suggesting a threshold effect for extreme obesity [6]. Potential mechanisms include increased fat deposition in the neck and pharynx, further reductions in FRC, and higher prevalence of comorbidities such as obesity hypoventilation syndrome. Nonetheless, studies in elective settings remain inconclusive; for example, Mahmoud et al. found that neither super-obesity nor super-super-obesity independently predicted difficult intubation or mask ventilation, with high STOP-Bang and Mallampati scores emerging as the primary predictors.

Critically ill patients differ substantially from elective surgical populations, presenting with limited FRC, rapid desaturation during apnea, hemodynamic instability, and multiple comorbidities, which may amplify the impact of morbid and super obesity on peri-intubation outcomes. Consequently, the independent effect of BMI ≥40 kg/m² on peri-intubation complications in the ICU remains uncertain.

To address this knowledge gap, the present study was designed as the first investigation in the literature to directly compare peri-intubation adverse events between morbidly obese and super obese critically ill trauma patients.The partipicants hypothesize that super obese patients experience a higher incidence of severe peri-intubation complications compared with their morbidly obese counterparts, thereby providing novel insight into risk stratification and airway management in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≥40
* Admission to the surgical ICU and intubated during ICU stay
* Availability of complete clinical data

Exclusion Criteria:

* Age < 18 years
* BMI<40
* No intubation
* Incomplete or missing medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult trauma patients aged 18 years and older admitted to the surgical ICU at UF Health Jacksonville between January 1, 2023, and November 1, 2025, who had a BMI ≥40 kg/m² and underwent intubation
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Severe hypoxemia | 30 minutes
  SpO₂ <80% during intubation

SECONDARY OUTCOMES:
Major peri-intubation complications | 30 minutes
  Severe hypotension
hospital mortality | 28 days
  rate of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ayten SARAÇOĞLU, Prof,MD, Study Director — Florida University Jacksonville

IPD SHARING:
Plan to Share IPD: No